CLINICAL TRIAL: NCT06180395
Title: Relation Between Bone Mineral Density, Gross Motor Function and Quality of Life In Children With Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Talaat Elsayed Emara, Principal Investigator, Cairo University
Other Study IDs: CairoU_STE
Record Dates: First submitted 2023-12-05; First posted 2023-12-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Bone Density, Low; Gross Motor Development Delay
MeSH Terms: conditions — Cerebral Palsy; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Ambulant ): consisted of 37 children with CP classified to level I, II and III according to GMFCS., then:
  1. Dual-energy X-ray absorptiometry (DXA) scans will be used to assess bone mineral density (BMD).
  2. Gross motor function measurement scale (GMFM) will be used to assess gross motor function.
  3. Quality of Life Questionnaire for Children (CP QOL-Child) will be used to assess quality of life (QOL).
  Interventions: Other: Group 1
- Group 2 (Non-Ambulant ): consisted of 38 children with CP classified to level IV and V according to GMFCS.then:
  1. Dual-energy X-ray absorptiometry (DXA) scans will be used to assess bone mineral density (BMD).
  2. Gross motor function measurement scale (GMFM) will be used to assess gross motor function.
  3. Quality of Life Questionnaire for Children (CP QOL-Child) will be used to assess quality of life (QOL).
  Interventions: Other: Group 2

INTERVENTIONS:
Other: Group 1 — consisted of 37 children with CP classified to level I, II and III according to GMFCS., then:
  Dual-energy X-ray absorptiometry (DXA) scans will be used to assess bone mineral density (BMD).
  Gross motor function measurement scale (GMFM) will be used to assess gross motor function.
  Quality of Life Questionnaire for Children (CP QOL-Child) will be used to assess quality of life (QOL).
  Other Names: Ambulant
  Groups: Group 1 (Ambulant )
Other: Group 2 — consisted of 38 children with CP classified to level IV and V according to GMFCS. then:
  Dual-energy X-ray absorptiometry (DXA) scans will be used to assess bone mineral density (BMD).
  Gross motor function measurement scale (GMFM) will be used to assess gross motor function.
  Quality of Life Questionnaire for Children (CP QOL-Child) will be used to assess quality of life (QOL).
  Other Names: Non-Ambulant
  Groups: Group 2 (Non-Ambulant )

SUMMARY:
studying the relationship between Bone Mineral Density, Gross Motor Function and, Quality of Life with CP can provide valuable insights into the musculoskeletal consequences of motor impairments and guide interventions to improve bone health.

Statement of the problem Is there a relation between Bone Mineral Density, Gross Motor Function and Quality of Life in children with CP ? Purpose of the study

To study the relationship between:

1. Bone Mineral Density and Gross Motor Function in ambulant and non-ambulant CP children.
2. Bone Mineral Density and Quality of Life in ambulant and non-ambulant CP children.
3. Gross Motor Function and Quality of Life in ambulant and non-ambulant CP children.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is primarily a neuromotor disorder that affects the development of movement, muscle tone and posture. The underlying pathophysiology is an injury to the developing brain in the prenatal through neonatal period. Although the initial neuro pathologic lesion is non-progressive, children with cerebral palsy may develop a range of secondary conditions over time that will variably affect their functional abilities. The prevalence of CP varies between 1.5 to more than 4 cases per 1,000 live births worldwide. The motor impairments associated with CP can range from mild to severe, affecting different muscle groups and leading to difficulties in activities of daily living and participation in social and recreational activities.

Children with CP often experience motor impairments that affect their gross motor function, leading to limitations in activities and participation. These motor impairments can also have a negative impact on bone health, resulting in reduced bone mineral density (BMD) and increased risk of skeletal complications.

Gross motor function (GMF) refers to the ability to perform coordinated movements using large muscle groups, such as walking, running, and jumping. It is a key aspect of physical ability and independence in daily activities for children with CP. Previous research has shown that gross motor function is closely associated with bone health in this population. However, further investigation is needed to explore the specific nature of this correlation and its implications for intervention strategies.

Gross motor function is commonly assessed using standardized tools such as the Gross Motor Function Classification System (GMFCS) or the Gross Motor Function Measure (GMFM). Quality of life is a multidimensional construct that encompasses physical, psychological, and social well-being. In the context of cerebral palsy, understanding the impact of gross motor function on quality of life is crucial for comprehensive care and intervention planning. Children with CP may face limitations in mobility, participation in activities, and social interactions, which can significantly affect their overall quality of life. Exploring the relationship between gross motor function and quality of life can provide valuable insights into the factors influencing the holistic well-being of children with CP.

The quality of life in children with CP is not only influenced by their motor function but also by their overall health and well-being. Bone health plays a crucial role in maintaining the physical abilities and independence of individuals, as well as their overall quality of life. Impaired bone health in children with CP can lead to limitations in mobility, increased pain, and reduced participation in activities, which can have a significant impact on their overall well-being.

Bone mineral density, on the other hand, is an important measure of bone strength and overall skeletal health. Children with CP often exhibit lower BMD compared to typically developing peers due to factors such as reduced weight-bearing activities, muscle weakness, altered biomechanics, limited mobility, and hormonal imbalances. This reduced BMD increases their susceptibility to fractures and skeletal deformities, further impacting their functional abilities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Children with CP (spastic diplegia and quadriplegia).
2. Their chronological ages will be ranged from 7 to 10 years.
3. They will be selected from both genders.
4. Their motor function will be at any Level according to GMFCS.
5. Their body mass index (BMI ) will be normal.

Exclusion criteria

Children will be excluded from the study if they have any of the following :

1. Underweight, Overweight or Obese.
2. Epilepsy , kidney problems that make them taking hormonal treatments or drugs affect bone density or taking calcium, vitamin D, steroids during 6 months prior to the study.
3. Fracture in the measurement areas.
4. Hip Flexion deformity more than 30° when posed to measure.
5. Internal metallic fixations in the measurement areas (neck of femur and lumber vertebra from L1-L4).
6. Hyperthyroidism or Hypothyroidism.
7. Hypotonia.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Seventy- five CP Children will be divided into two groups according to GMFCS:
  1. Group 1 (Ambulant ) consisted of 35 children with CP classified to level I, II and III according to GMFCS.
  2. Group 2 (Non-Ambulant ) consisted of 35 children with CP classified to level IV and V according to GMFCS.
  All measured variables will be identified for children of both groups, then correlation between BMD, gross motor function and QoL will be determined.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry (DXA) scans | 1 day
  Dual-energy X-ray absorptiometry (DXA) scans will be used to assess bone mineral density (BMD).
Gross motor function measurement scale (GMFM) | 1 day
  Gross motor function measurement scale (GMFM) will be used to assess gross motor function.
Quality of Life Questionnaire for Children (CP QOL-Child) | 1 day
  Quality of Life Questionnaire for Children (CP QOL-Child) will be used to assess quality of life (QOL).

CONTACTS AND LOCATIONS:
Overall Officials: Elham Elsayed Salem, professor, Study Chair — Cairo University
Locations (1):
- faculty of medicine , Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP